CLINICAL TRIAL: NCT03261921
Title: Adjuncts to Caudal Block in Pediatrics
Brief Title: Caudal Combination of Dexamethasone and/or Dexmedetomidine to Bupivacaine in Pediatric Hypospadias Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amany Hassan Saleh, principal investigator,MD of anesthesia and intensive care unit., Cairo University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Diagnostic
Other Study IDs: N-43-2016
Record Dates: First submitted 2017-08-07; First posted 2017-08-25 (Actual); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Caudal Block
MeSH Terms: interventions — Dexamethasone; Calcium Dobesilate; Dexmedetomidine; Bupivacaine

STUDY DESIGN:
Intervention Model Description: Sixty-three patients with ASA I-II aged from 1-6 years scheduled for hypospadias surgery in Abu El-Resh pediatric Hospital-Cairo university, were included in this prospective randomized double-blinded clinical study. Patients with contraindication to caudal anesthesia, cardiovascular diseases, drug allergy, type I diabetes, clotting disorders, mentally retarded children or those whose families did not approve inclusion in the study were excluded from the study.
  Patients were randomly divided on the morning of surgery into three groups group I( dexamethasone 21 patients), Group II ( Dexmedetomidine 21 patients) and group III(Dexmedetomidine and dexamethasone 21 patients).
Who Masked: Participant, Care Provider, Investigator
Masking Description: The Patients allocated to study groups using computer generated random list & group assignment was sealed in sequentially numbered opaque envelopes that opened after induction of anesthesia.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dexamethasone group (Active Comparator): In this group the patients received 0.5 ml/kg of bupivacaine 0.25% + (0.1 mg/kg dexamethazone) caudally.
  Interventions: Drug: Dexamethasone; Drug: Bupivacaine
- Dexmedetomidine group (Active Comparator): In this group the Patients received 0.5 ml/kg of bupivacaine 0.25% + dexmedetomidine(1 mu/kg) caudally.
  Interventions: Drug: Dexmedetomidine; Drug: Bupivacaine
- Combination group (Active Comparator): In this group the patients received 0.5 ml/kg of bupivacaine 0.25% + dexamethasone(0.1mg/kg) and dexmedetomidine (1 mu/kg) caudally.
  Interventions: Drug: Dexamethasone; Drug: Dexmedetomidine; Drug: Bupivacaine

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone is used peri -operatively mainly to prevent nausea and vomiting. Also epidural administration of dexamethasone prolong the postoperative analgesia and reduce analgesic needs
  Other Names: decadron
  Arms: Combination group; Dexamethasone group
Drug: Dexmedetomidine — Dexmedetomidine is an alpha 2 agonist which has sedative ,analgesic, opioid sparing effect and was proved to prolong the duration of postoperative analgesia when added to local anesthetics
  Other Names: precedex
  Arms: Combination group; Dexmedetomidine group
Drug: Bupivacaine — local anesthetic agent
  Other Names: plain marcaine

SUMMARY:
One of the most commonly used regional anesthetic techniques in pediatric surgeries is the caudal epidural block. Its main disadvantage remains the short duration of action. Hence, different additives have been used. Dexmedetomidine as an additive to the local anesthetic bupivacaine in caudal epidural analgesia prolongs the duration of postoperative analgesia so is dexamethasone. The investigators aimed to study the effect of combining both additives in the duration of analgesia, decreasing side effects and decreasing anesthetic doses

DETAILED DESCRIPTION:
Sixty three children scheduled for hypospadias randomized into 3 groups. Group I (n=21) (dexamethasone 0.1mg/kg+ 0.5ml/kg bupivacaine 0.25%), group II(n=21)( dexmedetomidine 0.01ug/kg+ 0.5ml/kg bupivacaine 0.25%)and groupIII(n=21)(dexamethasone0.1mg/kg+dexmedetomidine0.01ug/kg +0.5ml/kg bupivacaine 0.25%).intraoperative and postoperative hemodynamics were recorded. In PACU, MOPS scores and sedation scores were recorded at 30min,1,2,3,6and 12hrs. Also the time of first analgesic request was recorded.

ELIGIBILITY:
Inclusion Criteria:

1 - ASA I-II 2- Males only 3- Children aged from 1-6 years 4- Children scheduled for hypospadias surgery

Exclusion Criteria:

1. Contraindication to caudal anesthesia.
2. cardiovascular diseases.
3. drug allergy.
4. Type I diabetes.
5. Clotting disorders.
6. Mentally retarded children or those whose families did not approve inclusion in the study

Ages: 1 Year to 6 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — males candidate for hypospadias surgery
Enrollment: 63 (Actual)
Dates: Start 2016-06-05 (Actual); Primary Completion 2017-06-22 (Actual); Study Completion 2017-07-07 (Actual)

PRIMARY OUTCOMES:
Time of first request of analgesia | 12 hours
  the time from caudal block to the first time to analgesic needs
pain scores | 12 hours
  the modified objective pain score

SECONDARY OUTCOMES:
sedation score | 12 hours
  ramsay sedation score at the time of pain
heart rates(beat/minute) | 3 hours.
  Intra-operative recording
mean arterial pressure (mmhg) | 3 hours
  Intra-operative recording

IPD SHARING:
Plan to Share IPD: No